CLINICAL TRIAL: NCT02384278
Title: Internet Based Cognitive Behavior Treatment for Alcohol Problems: A Pilot Study
Brief Title: Internet Based Cognitive Behavior Treatment for Alcohol Problems
Acronym: ICBT-AP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Anne H Berman, Associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID10
Record Dates: First submitted 2015-02-26; First posted 2015-03-10 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Alcohol Use Disorders
Keywords: alcohol use disorder; internet; cognitive behavior therapy; relapse prevention
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Internet-based CBT for alcohol problems (Experimental): A 12-week internet-based cognitive behavior treatment (CBT) and relapse prevention program. The subjects will have access to a psychologist guiding them through the program.
  Interventions: Behavioral: Internet-based CBT for alcohol problems

INTERVENTIONS:
Behavioral: Internet-based CBT for alcohol problems — A 12-week internet-based program based on cognitive behavior treatment (CBT) and relapse prevention

SUMMARY:
The purpose of this study is to determine whether internet based cognitive behavior therapy might be effective in the treatment of alcohol problems.

DETAILED DESCRIPTION:
A 12 week Internet based self help program based on cognitive behavioral therapy and relapse prevention is tested among Internet help seekers as well as among patients seeking help in addiction care.The design is a one armed pilot study, and outcomes are measured in terms of changes in alcohol consumption, problematic alcohol use, self efficacy, craving, as well as depression and quality of life. 20 participants are recruited entirely online from an open access website and 20 participants are recruited through information given to them at an addiction clinic. All participants have access to the same self help program and have access to a licensed psychologist who guides the person all the way through the program.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* access to the Internet
* problematic alcohol use defined as ≥ 16 p or more for men and ≥ 14 p or more for women in the Alcohol Use Identification Scale

Exclusion Criteria:

* not adequately fluent in Swedish
* reading or writing impairment if this is so severe as to affect treatment
* ongoing psychological treatment with content similar to the treatment being studied
* suicide risk defined as ≥ 4 p på MADRS-S Q 9 or through a telephone interview with clinician
* severe depression defined as MADRS-S ≥ 30 p
* somatic or psychiatric conditions that are contraindicated for the treatment such as psychosis, bipolar disorder (depressive or manic phase), severe post traumatic stress disorder.
* has during the last 3 weeks begun using medication for alcohol problems or other psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Time Line Follow Back (TLFB) | Baseline, 14 and 26 weeks
  Change in total TLFB score (consumption during preceding week), as a summarized

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT) | Baseline, 14 and 26 weeks
  Change in total AUDIT score, as a summarized measure of alcohol use (including alcohol consumption and alcohol-related problems)
Drug Use Identification Test (DUDIT) | Baseline, 14 and 26 weeks
  Change in total DUDIT score, as a summarized measure of drug use (including drug consumption and drug-related problems)
Montgomery Asberg Depression Rating Scale - self report (MADRS-S) | Baseline, 14 and 26 weeks
  Change in total MADRS-S score, as a summarized measure of depression
World Health Organization Quality of Life Scale (WHOQOL-BREF) | Baseline, 14 and 26 weeks
  Change in total WHOQOL-BREF score, as a summarized measure of quality of life
Alcohol Abstinence Self Efficacy Scale (AASES) | Baseline, 14 and 26 weeks
  Change in total AASES score, as a summarized measure of self efficacy
Penn Alcohol Craving Scale (PACS) | Baseline, 14 and 26 weeks
Readiness to Change Questionnaire (RTCQ) | Baseline, 14 and 26 weeks
  Score in RTCQ as a summarized measure of motivation used as predictor for other outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Berman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institutet, Department of Clinical Neuroscience, Center for Psychiatric Research, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The dataset, unidentified, with background characteristics and outcomes is available as below.
Supporting Information: ICF
Time Frame: Since January 31, 2017
Access Criteria: Availability of data and materials
  The data set supporting the results of this article is available in the Open ICPSR repository with the following identifying information: Berman, A. H. (2017-01-31). High-intensity therapist-guided internet-based cognitive behavior therapy for alcohol use disorders - a pilot study. [Data set]. Ann Arbor, MI:
  Inter-university Consortium of Political and Social Research [distributor]. http://doi.org/10.3886/E100415V1.
URL: http://doi.org/10.3886/E100415V1

REFERENCES:
- [Derived] Sundstrom C, Kraepelien M, Eek N, Fahlke C, Kaldo V, Berman AH. High-intensity therapist-guided internet-based cognitive behavior therapy for alcohol use disorder: a pilot study. BMC Psychiatry. 2017 May 26;17(1):197. doi: 10.1186/s12888-017-1355-6. PMID 28549424